CLINICAL TRIAL: NCT04071561
Title: Prevention of Conversion in Posterior Retroperitoneal Adrenalectomy by Measuring Preoperative Anatomical Conditions on Cross-sectional Imaging (CT or MRI)
Brief Title: Prevention of Conversion in Posterior Retroperitoneal Adrenalectomy by Measuring Preoperative Anatomical Conditions
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Collaborators: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Simone Eichelberger, BMed, University of Basel
Other Study IDs: 201901147
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Adrenal Tumor; Adrenal Mass; Pheochromocytoma; Conn Adenoma; Adrenal Metastases; Adrenal Hyperplasia
Keywords: Adrenalectomy; Minimally invasive surgery; Posterior Retroperitoneoscopic adrenalectomy; Retroperitoneal fat mass
MeSH Terms: conditions — Adrenal Gland Neoplasms; Pheochromocytoma; Adrenocortical Adenoma; Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-conversion: In 13 patients, 14 posterior retroperitoneal adrenalectomy procedures were successfully completed and form the non-conversion group
  Interventions: Other: Posterior retroperitoneal adrenalectomy (PRA)
- Conversion: Conversion to lateral transperitoneal adrenalectomy was necessary in 1 patient after starting posterior retroperitoneal adrenalectomy.
  Interventions: Other: Posterior retroperitoneal adrenalectomy (PRA); Other: Lateral transperitoneal adrenalectomy (LTA)

INTERVENTIONS:
Other: Posterior retroperitoneal adrenalectomy (PRA) — Minimally invasive adrenalectomy procedure
Other: Lateral transperitoneal adrenalectomy (LTA) — During posterior retroperitoneal adrenalectomy, the failure to progress or the difficulty of creating or maintaining a pneumoperitoneum are reasons why conversion occurs.
  Groups: Conversion

SUMMARY:
With our retrospective study the investigators show the limitations of the posterior retroperitoneal adrenalectomy by analyzing anatomical parameters.

The investigators compared the data from one patient who underwent a conversion with 13 patients without a conversion. Furthermore, they explored the influence of these parameters on the operation time and excluded the patient who had a conversion from this analysis.

The investigators hypothesize that by determining anatomical characteristics on cross-sectional imaging (CT or MRI), they can show the limitations of the posterior retroperitoneal adrenalectomy to prevent patients from being converted to lateral transperitoneal adrenalectomy.

DETAILED DESCRIPTION:
Minimally invasive adrenalectomy has become the gold standard for the surgical treatment of small, benign adrenal lesions. In addition to the common laparoscopic lateral transperitoneal adrenalectomy, the posterior retroperitoneal adrenalectomy is becoming increasingly important.

To date, there is no consensus regarding the preferred approach in the resection of benign adrenal tumors. A comprehensive adrenal tumor program should be able to offer both options, however, patient selection criteria for a given approach have not yet been defined. The choice between lateral transperitoneal adrenalectomy and posterior retroperitoneal adrenalectomy is relevant for patients with unilateral tumors < 6-7 cm and without previous abdominal surgery.

The aim of this study was to determine the limits of posterior retroperitoneal adrenalectomy using anatomical parameters to enable the preferred access to be chosen preoperatively to prevent conversion. In addition, the investigators describe the relationship between these parameters and the operation time to find a measure of the degree of technical difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose adrenal gland was removed with retroperitoneal access
* Operation was between 01.07.2016 and 31.12.2018
* Operation was at the Kantonsspital Aarau

Exclusion Criteria:

* Patients with multivisceral resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent posterior retroperitoneal adrenalectomy at Kantonsspital Aarau.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Sagittal distance between the dorsal border of the adrenal gland and the 12th rib tip | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Sagittal distance between the dorsal border of the adrenal gland and the 12th rib tip, mm.
Thickness of retroperitoneal fat | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Defined as the largest distance between the kidney parenchyma and the posterior abdominal wall at the level where the renal vein joins the vena cava inferior.
Posterior Adiposity Index | The measurement of the parameter from the cross-sectional image was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Distance from skin to renal parenchyma through the 12th rib tip. The larger the distance, the larger the index. The scale ranges are open.
Longitudinal distance between the upper pole of the kidney and the inferior border of the adrenal gland. | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Longitudinal distance between the upper pole of the kidney and the inferior border of the adrenal gland, mm.
Longitudinal distance between the superior border of the adrenal gland to the 12th rib tip. | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Longitudinal distance between the superior border of the adrenal gland to the 12th rib tip, mm.
Longitudinal distance between the 12th rib and the iliac crest | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Longitudinal distance between the 12th rib and the iliac crest, mm.
Sagittal thickness of the subcutaneous layer above the 12th rib tip | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Sagittal thickness of the subcutaneous layer above the 12th rib tip, mm.
Sagittal thickness of the subcutaneous layer above the iliac crest | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Sagittal thickness of the subcutaneous layer above the iliac crest, mm.
Thickness of the subcutaneous layer above the 12th rib tip | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Thickness of the subcutaneous layer above the 12th rib tip, measured on the straight line to the center of gravity, mm.
Sagittal thickness of the subcutaneous layer between the center of gravity and the lateral border of the body | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Sagittal thickness of the subcutaneous layer between the center of gravity and the lateral border of the body, measured at the level of the 12th rib tip, mm.
Tumor size | The measurement was performed in the period from 19.11.2018 - 04.02.2019.
  Measurement of preoperative anatomical conditions on cross- sectional imaging (CT or MRI). Tumor size, cm.
Operative time | The data were collected between 19.11.2018 and 04.02.2019.
  Duration of adrenalectomy. Data were extracted and analyzed from the hospital information system.

SECONDARY OUTCOMES:
Body-Mass-Index | The data were collected between 19.11.2018 and 04.02.2019.
  Value derived from the mass (weight) and height of a person. Data were extracted and analyzed from the hospital information system.
The side of the adrenal gland that was removed | The data were collected between 19.11.2018 and 04.02.2019.
  Side of the removed adrenal gland (left, right, bilateral). Data were extracted and analyzed from the hospital information system.
Previously performed abdominal surgeries taken from the hospital information system | The data were collected between 19.11.2018 and 04.02.2019.
  Previous abdominal operations with opening of the abdominal cavity which give an indication of adhesions.Data were extracted and analyzed from the hospital information system.
Age | The data were collected between 19.11.2018 and 04.02.2019.
  Age at adrenalectomy. Data were extracted and analyzed from the hospital information system.
Sex | The data were collected between 19.11.2018 and 04.02.2019.
  Female or Male
Histological diagnosis of the sample from the adrenalectomy | The data were collected between 19.11.2018 and 04.02.2019.
  Histological evaluation. Data were extracted and analyzed from the hospital information system.
Imaging | The data were collected between 19.11.2018 and 04.02.2019.
  CT or MRI

CONTACTS AND LOCATIONS:
Overall Officials: Christian A Nebiker, PD Dr. med., Principal Investigator — Kantonsspital Aarau
Locations (1):
- Simone Eichelberger, Basel, Switzerland